CLINICAL TRIAL: NCT03634007
Title: A 52-Week, Multicenter, Phase 1/2 Open-label Study to Evaluate the Safety of LX1001 in Participants With APOE4 Homozygote Alzheimer's Disease
Brief Title: Gene Therapy for APOE4 Homozygote of Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lexeo Therapeutics (Industry)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LX1001-01
Record Dates: First submitted 2018-08-03; First posted 2018-08-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Early Onset Alzheimer Disease
Keywords: Alzheimer Disease; APOE4 homozygotes
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: 1.4 x 10^10 gc/mL CSF (Experimental): Participants will receive 1.4 x 10^10 gc/mL CSF of LX1001.
  Interventions: Biological: LX1001
- Cohort 2: 4.4 x 10^10 gc/mL CSF (Experimental): Participants will receive 4.4 x 10^10 gc/mL CSF of LX1001.
  Interventions: Biological: LX1001
- Cohort 3: 1.4 x 10^11 gc/mL CSF (Experimental): Participants will receive 1.4 x 10^11 gc/mL CSF of LX1001.
  Interventions: Biological: LX1001
- Cohort 4: 1.4 x 10^14 gc (fixed dose) (Experimental): Participants will receive 1.4 x 10^14 gc (fixed dose; approximately 3.4 × 10^11 gc/mL CSF based on an average CSF volume of 409 mL) of LX1001.
  Interventions: Biological: LX1001

INTERVENTIONS:
Biological: LX1001 — LX1001 is a serotype rh.10 AAV gene transfer vector expressing the cDNA coding for human APOE2.
  Other Names: AAVrh.10hAPOE2

SUMMARY:
This clinical trial is an open label, dose-ranging study designed to evaluate gene therapy to treat patients who are APOE4 homozygotes with clinical diagnosis varying from mild cognitive impairment due to Alzheimer's, mild dementia due to Alzheimer's disease, and moderate dementia due to Alzheimer's disease.

DETAILED DESCRIPTION:
The study will assess the safety and toxicity of intrathecal administration of AAVrh.10hAPOE2 (LX1001), serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the complementary deoxyribonucleic acid (cDNA) coding for human apolipoprotein E2 (APOE2), directly to the central nervous system (CNS)/ CSF of APOE4 homozygotes with Alzheimer's disease. All subjects will have evidence of cerebrospinal fluid (CSF) biomarkers consistent with Alzheimer's disease. The study will establish a maximum tolerable dose and generate preliminary evidence regarding whether direct administration of LX1001 to the CNS of those Alzheimer's patients will lead to conversion of the APOE protein isoforms in the CSF of APOE4 homozygotes from APOE4 to APOE2-APOE4.

ELIGIBILITY:
Inclusion Criteria:

* APOE4 homozygotes
* Willing and able to provide informed consent (or consent provided by a legally authorized representative)
* Clinical diagnosis of mild cognitive impairment due to Alzheimer's disease or mild to moderate dementia due to Alzheimer's disease
* Evidence of CSF biomarkers consistent with Alzheimer's disease
* Serum neutralizing anti-AAVrh10 titer <1:100
* No evidence of active infection of any type, including hepatitis virus (A, B, or C) or human immunodeficiency virus (HIV-1 and HIV-2)
* Fertile or infertile individuals; it will be recommended that fertile individuals utilize barrier birth control measures to prevent pregnancy for the duration of the study
* Individuals not receiving experimental medications or participating in another experimental protocol for at least 4 weeks prior to entry into the study
* Participants who agree not to post their personal data related to the study on social media.

Exclusion Criteria:

* Individuals receiving systemic immunosuppressant or corticosteroid therapy other than protocol-specified, are receiving a monoclonal anti-amyloid therapy (example, Aduhelm™ (aducanumab), Leqembi™ (lecanemab-irmb) or unable to wash out from anti-coagulant medications.
* Individuals who do not fit the American Journal of Neuroradiology recommendations for image-guided spinal procedures
* Presence of other significant medical, psychiatric, or neurological conditions may disqualify the participant from participation in this study, particularly those which would create an unacceptable risk of receiving the LX1001-01 vector, for example, malignancy, heart failure, liver or renal failure, or HIV positive.
* Elevated white blood cell count, temperature >38.5° C, infiltrate on chest x-ray. Note: Repeat of these examinations during the screening period is permitted to confirm eligibility
* Prior or concurrent participation in any gene and/or cell therapy
* Any condition, disorder, or abnormal laboratory test findings at screening which, in the judgment of the investigator, would interfere with the individual's ability to comply with all study requirements or would require the administration of treatment during the study that could potentially affect the interpretation of the study data, or would place the individual at unacceptable risk by his/her participation in the study
* Individuals who cannot participate in magnetic resonance imaging, amyloid and tau PET scans, and CSF studies
* Individuals who cannot undergo study-related procedures without general anesthesia (other than who need general anesthesia for the gene therapy administration)
* More than 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, or evidence of a prior macro hemorrhage on screening MRI
* Individuals with a history of clinically significant hypersensitivity or contraindication as judged by the investigator, to any component of the study drug formulation or to any drugs used in this study (examples are corticosteroids and proton-pump inhibitors)
* Are pregnant or nursing

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events and serious adverse events | 1 year
  Adverse events categorized and graded
The proportion of participants with treatment-emergent adverse events and serious adverse events at each dosage | 1 year
  Adverse events categorized and graded per study drug dose

CONTACTS AND LOCATIONS:
Overall Officials: Lexeo Clinical Trials, Study Director — Lexeo Therapeutics
Locations (4):
- United States (4):
  - K2 Medical Research, Maitland, Florida
  - PPD- Orlando Research Unit, Orlando, Florida
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De BP, Cram S, Lee H, Rosenberg JB, Sondhi D, Crystal RG, Kaminsky SM. Assessment of Residual Full-Length SV40 Large T Antigen in Clinical-Grade Adeno-Associated Virus Vectors Produced in 293T Cells. Hum Gene Ther. 2023 Aug;34(15-16):697-704. doi: 10.1089/hum.2023.032. PMID 37171121